CLINICAL TRIAL: NCT03457272
Title: Development and Evaluation of a Patient Safety Model Targeting Severe Clinical Deterioration and Safety Awareness in the Emergency Department
Brief Title: Development and Evaluation of a Patient Safety Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Horsens Hospital (Other); Central Jutland Regional Hospital (Other); Randers Regional Hospital (Other); Herning Hospital (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18296453
Record Dates: First submitted 2017-12-04; First posted 2018-03-07 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Emergency Medicine
Keywords: Patient Safety; Risk Factors; Quality Indicators, Health Care; Risk Assessment

STUDY DESIGN:
Intervention Model Description: The study consists of two intervention and two control departments. The intervention consists of a risk assesment to ensure systematic and standardized identification of patients in risk of clinical deterioration and a decision support algorithm. Actions are undertaken on the basis of the standardized decision support and when a patient is determined to be at risk escalation plans are activated. As part of the intervention, huddles are conducted and patients at risk are interdisciplinarily discussed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New risk assessment (Experimental): New risk assesment
  Interventions: Other: New risk assessment
- Standard (No Intervention): Standard risk assessment

INTERVENTIONS:
Other: New risk assessment — Consists of a simple physiological scoring system and an assessment of patients who should assist healthcare professionals in identifying patients at risk of clinical deterioration earlier and support timely response and escalation of observation, care and treatment and thereby prevent the development of severe clinical deterioration.
  The patients included in the study will be monitored using the new risk assessment tool with different intervals according to the patients' conditions. Underlying the tool are algorithms of action for intervention in the critically ill patient, inter professional guidelines and guidance for standardized monitoring, escalation plans and huddles.
  Arms: New risk assessment

SUMMARY:
Despite systems for early detection of critical illness, 12% of patients in the emergency department develop clinical deterioration with an increased risk of death as a result.

There is a need for a intervention to support the identification and clinical management of patients at risk of clinical deterioration earlier hospitalization. The Cincinnati Children's Hospital has introduced a model that systematically complements systems for early detection of critical illness with the assessment of patient and relatives concern, clinical intuition and concern of the staff. In addition, the model includes formalized organizational processes aimed at systematic review of risk patients and early treatment efforts. Studies from United States indicate that the model can lead to reduction of serious incidental events and increase the staff awareness of the situation. The Cincinnati model is designed for children and has not yet been studied in a controlled study.

Purpose To develop and investigate the impact of a Danish patient safety model. Method A literature review is conducted to identify risk factors that should be included in a model aimed at detecting and managing clinical deterioration. A patient safety model is developed on the basis of the literature review and the Cincinnati model and is tested in a pilot study. In a controlled intervention study, the effect is investigated against severe clinical deterioration. The intervention is carried out at the emergency departments at Horsens Regional Hospital and Viborg Regional Hospital with the regional hospitals in Randers and Herning as control departments.

DETAILED DESCRIPTION:
Preventing deterioration in acute patients is of great interest internationally. Studies demonstrate that clinical deterioration can be measured up to 24 hours before a heart arrest or intensive care admission in the vital signs. Therefore, the health services have implemented early warning systems to detect deterioration and critical illness.

Despite the systems, 12% of patients in an emergency department still develop severe clinical deterioration with increased risk of death as a result. Research indicates that the reasons for this may be diverse and further action to support the early identification and treatment of patients at risk of deterioration is needed.

Cincinnati Children's Hospital has introduced a patient safety model to ensure identification and mitigation of patient risk through escalated observation, care and treatment depending on the individual's risk for clinical deterioration. The model includes early warning systems, but as something new, it is supplemented with systematic evaluation of more subjective factors such as staff's clinical gaze and concerns, patient/relatives' concerns, communication problems and high risk therapy.

In an observational study, the Cincinnati Situation Awareness model was found to be associated with a near 50% reduction in unsafe intensive care unit transfers and decrease in severe safety events. However, the model has so far not been evaluated in a controlled study or an adult population.

The study will consist of three substudies; the overall study design is based on a framework for implementation of complex interventions following a four-step-process entailing development, pilot test, evaluation and reporting.

Study I. The study will consist of a systematic review and aims to identify risk factors associated with severe clinical deterioration and severe safety events that should ultimately be considered for inclusion in the patient safety model.

The aim of study II is to develop a patient safety model based on the components in the Cincinnati Situation Awareness model and explore its feasibility. The Danish patient safety model is expected to consist of systematic patient risk screening, bed huddles and audits of intensive care unit transfers.

Relevant aspects that should be included in the systematic patient risk screening are identified based on the literature study. A multidisciplinary panel is established to ensure that the choice of risk parameters is made on the basis of risk factors with the highest impact and the applicability to standard care.

A pilot test of the model will be conducted to evaluate the feasibility of methods and procedures based on the principles of the Medical Research Council guidance.

The final model will be investigated in a prospective controlled intervention study design to examine the effect in relation to severe clinical deterioration, safety awareness and serious adverse events (Study III).

The study will follow a Quasi-experimental design. The intervention will be implemented at the Emergency Departments and Intensive Care Units at Horsens and Viborg Regional Hospitals with the Emergency Departments at Herning and Randers Regional Hospitals as controls.

A positive outcome is expected to increase patient safety by reducing patients with severe deterioration, serious adverse events and increase staff safety awareness.

ELIGIBILITY:
Inclusion Criteria:

* Adult somatic patients (≥18 years) admitted to the participating Emergency Departments

Exclusion Criteria:

* Patients with injuries caused by trauma
* Patients received with cardiac arrest, as a surgical or medical call (can participate if admitted to the Emergency Department and not directly transferred to the Intensive Care Unit)
* Patients hospitalized with a psychiatric diagnosis as the primary cause of admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34556 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with severe clinical deterioration in the ED | Participants will be followed for the length of stay in the Emergency Department, an expected period of 48 hours
  Severe clinical deterioration will be measured by the early warning system used in Central Denmark Region based on vital signs collected from medical records. The score is aggregated and the vital signs include respiratory rate, SatO2, systolic blood pressure, pulse, temperature and level of consciousness measured by APVU.
  The initial deterioration process from score 0-1 will be considered as "no deterioration". Deterioration directly to score 2 and above, or deterioration from score ≥2 and further will be considered severe.

SECONDARY OUTCOMES:
Safety awareness | up to 4 weeks (in baseline and in intervention)
  Staff safety awareness will be measured in the last months of the baseline period and in the last months of the intervention period by the Safety Attitudes Questionnaire adapted and validated for Danish hospital settings. The questionnaire consists of 31 items rated on a 5-point Likert type scale. The questionnaire comprises six subscales: teamwork climate, safety climate, stress recognition, job satisfaction, working conditions, and perceptions of unit management.
Proportion of participants with severe safety events | Participants will be followed for the duration of the hospital stay in the Emergency Department, an expected average of 17 hours
  Severe safety events is a composite outcome consisting of either unexpected in-hospital cardiac/respiratory arrest, unexpected in-hospital death (when no Do-Not-Resuscitate order has been prescribed) and unanticipated intensive care unit transfer from the Emergency Department
Proportion of participants admitted to the Intensive Care Units from the Emergency Departments | Participants will be followed for the duration of the hospital stay in the Emergency Department, an expected average of 17 hours
  Proportion of participants referred to the Intensive Care Units from the Emergency Departments
Proportion of participants admitted to the Intensive Care Units from the wards | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  Proportion of participants admitted to the Intensive Care Units from the wards
Length of stay at the Intensive Care Unit | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  The length of time patients spend in the Intensive Care Units
Proportion of 30 day - readmission | Participants will be followed for the duration of 30 days after the hospital stay
  Readmission until 30 days after the Emergency Department admission (Central Denmark Region)
Length of stay in the Emergency Departments | Participants will be followed for the duration of the hospital stay in the Emergency Department, an expected average of 17 hours
  The length of time patients spend in the Emergency Department
Length of stay in the Hospital | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  The length of time patients spend in the hospital
Proportion of in-hospital death | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  The proportion of participants who die in the hospital
Proportion of in-hospital cardiac/respiratory arrest | Participants will be followed for the duration of hospital stay, an expected average of 1 week
  The proportion of participants who have a cardiac or respiratory arrest in the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Gitte B Tygesen, PhD student, Principal Investigator — Regionshospitalet Horsens
Locations (4):
- Denmark (4):
  - Herning Regional Hospital, Herning
  - Horsens Regional Hospital, Horsens
  - Randers Regional Hospital, Randers
  - Viborg Regional Hospital, Viborg